CLINICAL TRIAL: NCT00875381
Title: Immunohistochemical Analysis of Melanocytes in Sun-Exposed Skin
Brief Title: Analysis of Melanocytes (Pigment Cells) in Sun-Exposed Skin
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Lawrence E. Gibson, M.D., Mayo Clinic Rochester
Other Study IDs: 07-002038
Record Dates: First submitted 2009-04-02; First posted 2009-04-03 (Estimated); Last update posted 2011-03-15 (Estimated); Status verified 2011-03

CONDITIONS: Carcinoma, Basal Cell; Carcinoma, Squamous Cell
Keywords: Melanocytes
MeSH Terms: conditions — Carcinoma, Basal Cell; Carcinoma, Squamous Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The proposed dog-ears excised, that were to be discarded during reconstruction, were evaluated for the presence of any visible lesions (i.e. ephelid, lentigo, seborrheic keratosis, nevi). Dog-ears with any skin lesions were excluded. The specimens were inked by the surgeon on the side to be cut by the histotechnician. The specimens were placed in formalin bottles and submitted to the pathology department at Mayo Clinic Rochester for processing. The tissue was cut (4 microns) along its long access and stained with routine H& E and Mart-1 (MelanA) immunostains.
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to estimate and define the mean number, degree of confluence, and depth of penetration of melanocytes in chronically sun exposed skin of the head and neck using Mart-1 immunostains on frozen sections. The study was conducted to confirm whether similar results were found using permanent sections. The present study used hematoxaline and eosin (H&E) staining as well as Mart-1 staining, and included patients from both Mayo Clinic Jacksonville and Rochester.

DETAILED DESCRIPTION:
For each study participant we recorded their age, sex, state they lived in, tumor type, tumor location, recent sun exposure (during the two weeks prior to the surgery), whether or not a follicle was present on the slide, and if so the follicular extension (mm) from the granular layer, presence of atypia, nesting, pagetoid spread. Two slides were obtained; one stained with Mart-1; the other with H&E. For both, melanocyte counts per high power field (400 X HPF magnification) were obtained in three locations of the slide. The mean of the 3 counts was used for analysis, though the individual counts were considered in some data summaries (see below). Classification of photo-aging according to the Glogau scale was noted by the surgeon as type1: "no wrinkles"; type II "wrinkles in motion"; type III "wrinkles at rest" and type IV "only wrinkles." Confluence was categorized by the number of adjacent melanocytes as none, mild (2 side-by-side), moderate (3-6), or severe (7 or more).

ELIGIBILITY:
Inclusion Criteria:

* Participants undergoing Mohs and reconstructive surgery for basal cell and squamous cell carcinoma of the face and neck

Exclusion Criteria:

* Participants with a history of radiation to the head and neck were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 50 patients from Mayo Clinic Jacksonville and 50 Mayo Clinic Rochester will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2007-09; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
The mean number of melanocytes per high power field for Mart-1 was 12.7 in FL and 11.2 in MN. Using H&E, the means were 10.3 and 8.3 for FL and MN respectively. | one year

SECONDARY OUTCOMES:
Evidence of higher means in FL than in MN after adjusting for age and gender (p<0.001 for H&E, p=0.08 for Mart-1) and strong evidence of an increase in observed numbers of melanocytes with use of the Mart-1 stain compared to the H&E stain (p<0.001) | one year

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence E Gibson, MD, Principal Investigator — Mayo Clinic